CLINICAL TRIAL: NCT02233712
Title: An Open-label, Dose-finding, Schedule-changing, Multi-center Study to Determine the Antibody Response to G17DT Treatment of Patients With Gastric Cancer.
Brief Title: Open-label, Dose-finding Study to Determine Antibody Response to G17DT Treatment in Patients With Gastric Cancer.
Acronym: GC3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Advances Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC3
Record Dates: First submitted 2014-08-27; First posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Gastric Cancer
Keywords: gastric cancer, stomach neoplasms,
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): G17DT; 250 µg dose administered at 0, 1, and 3 weeks.
  Interventions: Biological: G17DT
- Group 2 (Experimental): G17DT; 100 µg dose administered at 0, 1, and 3 weeks.
  Interventions: Biological: G17DT
- Group 3 (Experimental): G17DT; 500 µg dose administered at 0, 1, and 3 weeks.
  Interventions: Biological: G17DT
- Group 4 (Experimental): G17DT; 500 µg dose administered at 0, 2, and 6 weeks.
  Interventions: Biological: G17DT

INTERVENTIONS:
Biological: G17DT
  Other Names: Polyclonal Antibody Stimulator (PAS)

SUMMARY:
An open label, dose-finding, schedule-changing, sequential, multiple dose, multi-center study in patients with Stage I-III gastric cancer. The first group of patients received a starting dose of 250 µg at weeks 0, 1, and 3. Thereafter, allocation to treatment with 100 µg or 500 µg was based on antibody response and dose tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed UICC Stage I, II or III gastric adenocarcinoma. Must have had a macroscopically curative resection for gastric cancer with absence of metastatic disease at the time of entry to the trial
* Male or female and over 18 years of age
* Must have a life expectancy of at least three months
* World Health Organization Performance Status of 0 to 1
* Given written conformed consent

Exclusion Criteria:

* Gastric surgery within four weeks of baseline (week 0) or gastric surgery anticipated in the period of the study
* History of other malignant disease within the previous five years, except non-melanomatous skin cancer or in situ carcinoma of the uterine cervix
* Previous use within the last four weeks, concomitant use or anticipated use in the period of the study, of any anti-cancer therapies
* Concomitant use of immunosuppressants, including systemic (i.e. oral or injected) corticosteroids
* Females who pregnant, planning to become pregnant or lactating
* Taking part in another study involving an investigational or licensed drug or device in the three months preceding enrollment or during this study
* Previously received G17DT treatment
* Haemoglobin (Hb) < 10.0 g/dL White blood cell count (WBC) < 4.0 x 10^9/L Platelets < 100 x 10^9/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 1999-08; Primary Completion 2000-03 (Actual)

PRIMARY OUTCOMES:
Antibody Levels | Up to Week 24
  Gastrin-17 antibodies are produced as a result of treatment with G17DT and the proportion of patients producing gastrin-17 antibodies was considered to be an appropriate measure of the immunogenicity of the dosing schedule under study.
Injection Site Reaction | Up to Week 12
  An examination was performed to assess injection site tolerability at every posttreatment visit from Week 1 to Week 12 (end of core phase).
World Health Organization (WHO) Performance Status | Up to Week 12
  WHO performance status was monitored up to Week 12 to compare final status with baseline status.
Diptheria Toxoid Antibody Levels | Up to Week 12
  Diptheria toxoid antibody levels were measured at screening and at Week 12 to assess toxicity from Diptheria toxoid.

SECONDARY OUTCOMES:
Adverse Events | Up to Week 24
  Any adverse events that were reported during the study

CONTACTS AND LOCATIONS:
Overall Officials: Peter G McCulloch, MB, ChB, Principal Investigator — University Hospital Aintree